CLINICAL TRIAL: NCT00813137
Title: A Multi-center Study of Folfox4 Combined With Recombinant Human Endostatin(Endostar)in Advanced Colorectal Cancer
Brief Title: FOLFOX4 Combined With Endostar in Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Collaborators: The Affiliated Changzhou Tumor Hospital of Suzhou University (Unknown)
Responsible Party: Yang Ling, the Affiliated Changzhou Tumor Hospital of Suzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: simcere0803
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-12

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Cancer; chemotherapy; recombinant human endostatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endostatins; endostar protein; Folfox protocol; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Folfox4 plus Endostar (Experimental)
  Interventions: Drug: Folfox4 plus recombinant human endostatin (Endostar)

INTERVENTIONS:
Drug: Folfox4 plus recombinant human endostatin (Endostar) — Endostar 15mg iv drip D1~7, D15~21, Oxaliplatin 85mg/m2 iv drip D1,15, CF 200mg/m2 iv drip D1,2,15,16, 5-Fu 400mg/m2 iv D1,2,15,16, 5-Fu 600mg/m2 civ D1,2,15,16
  Other Names: endostar; Folfox4; L-OHP; CF; 5-Fu

SUMMARY:
FOLFOX4 plus Avastin has been suggested as firstline regimen for advanced colorectal cancer by NCCN, a new angiogenesis inhibitor, known as Endostar(Recombinant Human Endostatin), prolonged the overall survival, time to progression and improved response rate in metastatic lung cancer in a large phase III clinical trial in china, so we design this trial to evaluate the safty and efficacy of FolFox4 plus Endostar in patients with advanced colorectal cancer

DETAILED DESCRIPTION:
Endostar is free supported by Shangdong Simcere Medgene biotech co.,Ltd. Endostar combination with Chemotherapy has been the first line treatment regimen to advanced NSCLC. Clinical data proved that Endostar was a wild spectrum and safe antiangiogenesis factor which could suppress almost 65 kinds of tumor mass in animal models and affect about 12 percent human genome. China NCCN colon or rectal cancer clinical practice guideline recommends Chemotherapy plus angiogenesis inhibitor as the first line treatment scheme. So we design FOLFOX4 plus Endostar to treat advanced colorectal cancer to research the RR and safety. We believe this treatment regimen may be a new approach to the advanced colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed metastatic CRC
* Measurable disease according to Response Criteria In Solid Tumours (RECIST)
* Performance Status 0 - 2 according to ECOG (Eastern Cooperative Oncology Group) Performance Status
* Age 18~75
* Life expectancy > 3 months
* Signed informed consent (IC)
* Adequate haematological and biological functions

Exclusion Criteria:

* Pregnant or lactating women
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs
* Neuropathy, brain, or leptomeningeal involvement
* Treatment with any biologic, cytotoxic, radiation , or hormonal therapy within four weeks.
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months or high risk/uncontrolled arrhythmia
* Uncontrolled significant comorbid conditions and previous radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Time to progression | every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Yang Ling, M.D, Ph.D, Principal Investigator — The Affiliated Changzhou Tumor Hospital of Suzhou University
Locations (2):
- China (2):
  - The Affiliated Changzhou Tumor Hospital of Suzhou University, Changzhou, Jiangsu
  - The Affiliated Zhongda Hospital of Southeast University, Nanjing, Jiangsu